CLINICAL TRIAL: NCT02167945
Title: An Open-Label, Multicenter Study to Evaluate Long-term Outcomes With ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 With or Without Ribavirin (RBV) in Adults With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection (TOPAZ-II)
Brief Title: A Study to Evaluate Long-term Outcomes Following Treatment With ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 With or Without Ribavirin (RBV) in Adults With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Acronym: TOPAZ-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-222
Record Dates: First submitted 2014-06-18; First posted 2014-06-19 (Estimated); Results first posted 2022-04-06 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Chronic Hepatitis C Virus (HCV) Infection Genotype 1
Keywords: Hepatitis C Genotype 1; Compensated Cirrhosis; Cirrhosis; Naïve; Hepatitis C; Hepatitis C Virus; Treatment-Experienced; Relapser; Null responder; Non responder
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Fibrosis | interventions — paritaprevir; ombitasvir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABT-450/r/ABT-267 plus ABT-333 with or without ribavirin (RBV) (Experimental): Participants with HCV GT1b without cirrhosis received the 3-DAA (ABT-450/ritonavir/ABT-267 and ABT-333) regimen: two 75 mg ABT-450/50 mg ritonavir/12.5 mg ABT-267 tablets taken orally every morning (QD) and one ABT-333 250 mg tablet taken orally twice a day (BID) for 12 weeks. Participants with HCV GT1a without cirrhosis and those with HCV GT1b with cirrhosis received the 3-DAA regimen and weight-based ribavirin (RBV; 1000 to 1200 mg divided twice daily per local label) for 12 weeks. Participants with HCV GT1a with cirrhosis received the 3-DAA regimen and weight-based RBV per local label for 24 weeks.
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: ABT-450/r/ABT-267 — Tablet for oral use
  Other Names: ABT-450 also known as paritaprevir; ABT-267 also known as ombitasvir; Paritaprevir/ritonavir/ombitasvir also known as Viekirax
Drug: ABT-333 — Tablet for oral use
  Other Names: ABT-333 also known as dasabuvir; ABT-333 also known as Exviera
Drug: Ribavirin (RBV) — Ribavirin was provided as 200 mg tablets, and dosed based on weight, 1000 to 1200 mg divided twice daily per local label. For example, for participants weighing < 75 kg, RBV may have been taken orally as 2 tablets in the morning and 3 tablets in the evening which corresponds to a 1000 mg total daily dose. For participants weighing ≥ 75 kg, RBV may have been taken orally as 3 tablets in the morning and 3 tablets in the evening which corresponds to a 1200 mg total daily dose.

SUMMARY:
The purpose of this study was to evaluate the effect of treatment with ABT-450 co-formulated with ritonavir and ABT-267 (ABT-450/r/ABT-267) and ABT-333; 3-DAA regimen, with or without ribavirin (RBV) in adults with chronic hepatitis C virus genotype 1 (HCV GT1) infection.

DETAILED DESCRIPTION:
This study (TOPAZ-II; M14-222), was a Phase 3b, open-label, multicenter study conducted in the United States which, together with its companion study TOPAZ-I (M14-423; NCT02219490) conducted outside of the United States, was designed with the primary objective of assessing the effect of treatment response on long-term clinical outcomes in adults with chronic HCV GT1 infection with or without compensated cirrhosis, who were either treatment-naïve or interferon/ribavirin (IFN/RBV) treatment- experienced. In both studies, participants were treated with the 3-DAA regimen with or without RBV. This study consisted of a screening period of up to 42 days, a treatment period of either 12 weeks for HCV GT1a-infected subjects without cirrhosis and for HCV GT1b-infected subjects without cirrhosis or with compensated cirrhosis or 24 weeks for GT1a-infected participants with compensated cirrhosis, and a 260-week post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Females must be post-menopausal for more than 2 years or surgically sterile or practicing specific forms of birth control
2. Chronic hepatitis C, genotype 1-infection (HCV RNA level greater than 1,000 IU/mL at screening)
3. HCV genotype 1 infection per screening laboratory result

Exclusion Criteria:

1. Use of contraindicated medications within 2 weeks of dosing
2. Abnormal laboratory tests
3. Positive hepatitis B surface antigen and anti-Human Immunodeficiency Virus Antibody
4. History of solid organ transplant, clinical evidence of Child-Pugh B or C classification or clinical history of liver decompensation
5. Presence of hepatocellular carcinoma at screening

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (48):
- United States (48):
  - St. Josephs Hospital and Med Center /ID# 127800, Phoenix, Arizona
  - Franco Felizarta, Md /Id# 126569, Bakersfield, California
  - Ruane Clinical Research Group /ID# 126577, Los Angeles, California
  - California Pacific Medical Center /ID# 128681, San Francisco, California
  - Univ of Colorado Cancer Center /ID# 126568, Aurora, Colorado
  - Medstar Health Research Institute /ID# 128683, Washington D.C., District of Columbia
  - Bach and Godofsky Infec Dis /ID# 128685, Bradenton, Florida
  - University of Florida - Archer /ID# 127787, Gainesville, Florida
  - Encore Borland-Groover Clinical Research /Id# 127781, Jacksonville, Florida
  - University of Miami /ID# 127622, Miami, Florida
  - South Florida Ctr Gastro, P.A. /ID# 126567, Wellington, Florida
  - Atlanta Gastro Assoc /ID# 126571, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 128684, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 126576, Chicago, Illinois
  - Duplicate_Indiana University Health /ID# 126573, Indianapolis, Indiana
  - Tulane University /ID# 127779, New Orleans, Louisiana
  - Louisana Research Center, LLC /ID# 126561, Shreveport, Louisiana
  - Johns Hopkins University /ID# 127791, Baltimore, Maryland
  - Digestive Disease Associates - Catonsville /ID# 127624, Catonsville, Maryland
  - Beth Israel Deaconess Medical Center /ID# 126560, Boston, Massachusetts
  - Henry Ford Health System /ID# 127783, Detroit, Michigan
  - Minnesota Gastroenterology PA /ID# 126579, Plymouth, Minnesota
  - St. Louis University /ID# 126564, St Louis, Missouri
  - AGA Clinical Research Associates, LLC /ID# 126578, Egg Harbor, New Jersey
  - Rutgers New Jersey School of Medicine /ID# 128686, Newark, New Jersey
  - University of New Mexico /ID# 128859, Albuquerque, New Mexico
  - Southwest Care Center /ID# 127784, Santa Fe, New Mexico
  - North Shore University Hospital /ID# 126565, New Hyde Park, New York
  - The Mount Sinai Hospital /ID# 128682, New York, New York
  - Columbia Univ Medical Center /ID# 126566, New York, New York
  - Columbia Univ Medical Center /ID# 127621, New York, New York
  - Premier Medical Group - GI Division /ID# 127793, Poughkeepsie, New York
  - Univ Rochester Med Ctr /ID# 127655, Rochester, New York
  - Atrium Health Carolinas Medical Center /ID# 127632, Charlotte, North Carolina
  - Carolinas Center For Liver Dis /ID# 127788, Statesville, North Carolina
  - University of Cincinnati Physicians Company, LLC /ID# 127790, Cincinnati, Ohio
  - Options Health Research, LLC /ID# 127630, Tulsa, Oklahoma
  - University Gastroenterology /ID# 127789, Providence, Rhode Island
  - Gastro One /ID# 127792, Germantown, Tennessee
  - Inquest Clinical Research /ID# 126574, Baytown, Texas
  - Cure C Consortium /ID# 126570, Houston, Texas
  - Liver Associates of Texas, P.A /ID# 126563, Houston, Texas
  - Austin Institute for Clinical Research /ID# 126562, Pflugerville, Texas
  - TX Liver Inst, Americ Res Corp /ID# 127623, San Antonio, Texas
  - Clinical Research Ctrs America /ID# 127780, Murray, Utah
  - Virginia Mason - Seattle Orthapedics /ID# 130288, Seattle, Washington
  - University of Washington /ID# 127785, Seattle, Washington
  - Dean Clinic /ID# 126575, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety population: All participants enrolled in this study (M14-222; TOPAZ-II) who received at least one dose of study drug
Period: Overall Study
Arm/Group | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV)
Started | 615
Completed | 366
Not Completed | 249
Not completed — Adverse Event | 16
Not completed — Withdrew Consent | 42
Not completed — Lost to Follow-up | 122
Not completed — COVID-19 logistical restrictions | 6
Not completed — Other, not specified | 63

BASELINE CHARACTERISTICS:
Population: Safety population: All participants enrolled in this study (M14-222; TOPAZ-II) who received at least one dose of study drug
Arm/Group | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV)
Number analyzed (Participants) | 615
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 243
  Male | 372
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 520
  Black or African American | 84
  Asian | 4
  American Indian or Alaska Native | 4
  Native Hawaiian or Other Pacific Islander | 0
  Multiple | 3
HCV Genotype 1 Subtype [Count of Participants; unit: Participants]
  GT1b without cirrhosis | 141
  GT1b with compensated cirrhosis | 22
  GT1 Non-b without cirrhosis | 359
  GT1 Non-b with compensated cirrhosis | 93
Prior HCV Treatment History [Count of Participants; unit: Participants]
  Treatment Naïve | 437
  Treatment Experienced | 178

OUTCOME MEASURES:

1. Primary Outcome: All-Cause Death: Time to Event
Description: Time to all-cause death was defined as the number of days from the first day of study drug dosing for the participant to the date of death. All deaths were to be included, regardless of whether the death occurred while the participant was still taking study drug or had previously discontinued study drug. If the participant did not die, their data was to be censored at the date of their last available assessment of clinical outcomes. For participants with no post-baseline assessment, the participant's data was to be censored on the first day of study drug dosing. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of all-cause death included pooled data from TOPAZ-II (this study) and the companion study TOPAZ-I (M14-423; NCT02219490).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: Intent-to-treat (ITT) population: all enrolled participants in this study (TOPAZ-II; M14-222; ITT-II) and in companion study M14-423 (TOPAZ-I; NCT02219490; ITT-I) who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12; Participants in Studies M14-222 and M14-423 Who Achieved SVR12: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ) 12 weeks after the last actual dose of study drug.
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 8.3 [3.1 to 21.2] | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 104 | 8.3 [3.1 to 21.2] | 0.7 [0.4 to 1.1]
  Kaplan-Meier estimate at PT Week 156 | 8.3 [3.1 to 21.2] | 1.2 [0.8 to 1.8]
  Kaplan-Meier estimate at PT Week 208 | 8.3 [3.1 to 21.2] | 1.5 [1.1 to 2.2]
  Kaplan-Meier estimate at PT Week 260 | 8.3 [3.1 to 21.2] | 2.0 [1.5 to 2.8]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; Comparisons between participants in studies M14-222 and M14-423 who achieved SVR12 and those who did not were performed using a log-rank test; Test type: Superiority; p < 0.001, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; A Cox proportional hazards (PH) model was constructed. The covariates for the model included baseline age, BMI, HCV genotype 1 subtype (1b, non-1b), IL28B genotype (CC, non-CC), prior treatment history (naive, experienced), baseline HCV RNA levels, baseline fibrosis stage (F0-1, F2, F3, F4), baseline albumin, baseline creatinine clearance, baseline platelet count, history of diabetes (yes, no), APRI, race (white, other), and alcohol use status (current, former, non-drinker); Test type: Superiority; p < 0.001, Cox proportional hazards model; Cox Proportional Hazard Ratio = 0.126, 95% CI 2-sided [0.044 to 0.358] — The estimated value represents the hazard ratio for developing the event in the group of participants in studies M14-222 and M14-423 who achieved SVR12 compared to the group of participants in studies M14-222 and M14-423 who didn't achieve SVR12

2. Primary Outcome: Liver-Related Death: Time to Event
Description: Time to liver-related death was defined as number of days from the 1st day of study drug dosing for the participant to date of liver-related death. All liver-related deaths were to be included, regardless of whether the death occurred while the participant was still taking study drug or had previously discontinued study drug. If the participant didn't experience the event of interest nor had died (all-cause death), their data was to be censored at the date of their last available assessment of clinical outcomes. For participants with no post-baseline assessment, their data was to be censored on the 1st day of study drug dosing. All-cause death was a censoring event for liver-related death. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of liver-related death included pooled data from TOPAZ-II (this study) and the companion study TOPAZ-I (M14-423; NCT02219490).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 1.4 [0.2 to 9.6] | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit
  Kaplan-Meier estimate at PT Week 104 | 1.4 [0.2 to 9.6] | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit
  Kaplan-Meier estimate at PT Week 156 | 1.4 [0.2 to 9.6] | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 208 | 1.4 [0.2 to 9.6] | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 260 | 1.4 [0.2 to 9.6] | 0.1 [0.1 to 0.4]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.007, Cox proportional hazards model; Cox Proportional Hazard Ratio = 0.031, 95% CI 2-sided [0.003 to 0.380] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Liver Decompensation: Time to Event
Description: Time to liver decompensation was defined as number of days from the 1st day of study drug dosing for the participant to the date of liver decompensation. All liver decompensation was to be included, regardless of whether it occurred while the participant was still taking study drug or had previously discontinued study drug. If the participant didn't experience the event of interest nor had died (all-cause death), their data was to be censored at the date of their last available assessment of clinical outcomes. For participants with no post-baseline assessment, their data was to be censored on the 1st day of study drug dosing. All-cause death was a censoring event for liver decompensation. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of liver decompensation included pooled data from TOPAZ-II (this study) and the companion study TOPAZ-I (M14-423; NCT02219490).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 4.5 [1.5 to 13.4] | 0.2 [0.1 to 0.5]
  Kaplan-Meier estimate at PT Week 104 | 4.5 [1.5 to 13.4] | 0.2 [0.1 to 0.5]
  Kaplan-Meier estimate at PT Week 156 | 4.5 [1.5 to 13.4] | 0.3 [0.1 to 0.6]
  Kaplan-Meier estimate at PT Week 208 | 4.5 [1.5 to 13.4] | 0.3 [0.2 to 0.7]
  Kaplan-Meier estimate at PT Week 260 | 4.5 [1.5 to 13.4] | 0.5 [0.2 to 0.9]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cox proportional hazards model; Cox Proportional Hazard Ratio = 0.038, 95% CI 2-sided [0.009 to 0.156] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Liver Transplantation: Time to Event
Description: Time to liver transplantation was defined as number of days from the 1st day of study drug dosing for the participant to date of liver transplantation. All liver transplantation was to be included, regardless of whether it occurred while the participant was still taking study drug or had previously discontinued study drug. If the participant didn't experience the event of interest nor had died (all-cause death), their data was to be censored at the date of their last available assessment of clinical outcomes. For participants with no post-baseline assessment, their data was to be censored on the 1st day of study drug dosing. All-cause death was a censoring event for liver transplantation. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of liver transplantation included pooled data from TOPAZ-II (this study) and the companion study TOPAZ-I (M14-423; NCT02219490).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit
  Kaplan-Meier estimate at PT Week 104 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit
  Kaplan-Meier estimate at PT Week 156 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 208 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 260 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.2 [0.1 to 0.5]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.860, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.997, Cox proportional hazards model — The Hazard Ratio for experiencing the event in the group of participants in studies M14-222 and M14-423 who achieved SVR12 compared to those who did not achieve SVR12 is infinite and the CI is not bounded due to zero events in one of the groups

5. Primary Outcome: Hepatocellular Carcinoma: Time to Event
Description: Time to hepatocellular carcinoma was defined as number of days from the 1st day of study drug dosing for the participant to date of hepatocellular carcinoma. All hepatocellular carcinoma was to be included, whether it occurred while the participant was still taking study drug or had previously discontinued study drug. If the participant didn't experience the event of interest nor had died (all-cause death), their data was to be censored at the date of their last available assessment of clinical outcomes. For those with no post-baseline assessment, their data was to be censored on the 1st day of study drug dosing. All-cause death was a censoring event for hepatocellular carcinoma. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of hepatocellular carcinoma included pooled data from TOPAZ-II (this study) and the companion study TOPAZ-I (M14-423; NCT02219490).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.2 [0.1 to 0.5]
  Kaplan-Meier estimate at PT Week 104 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.4 [0.2 to 0.8]
  Kaplan-Meier estimate at PT Week 156 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.5 [0.3 to 1.0]
  Kaplan-Meier estimate at PT Week 208 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.6 [0.4 to 1.1]
  Kaplan-Meier estimate at PT Week 260 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.9 [0.5 to 1.4]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.608, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.992, Cox proportional hazards model — [p-value comment as in outcome 4, analysis 2]

6. Primary Outcome: All-Cause Death, Liver-Related Death, Liver Decompensation, Liver Transplantation, Hepatocellular Carcinoma: Time to Event
Description: Time to the composite of clinical outcomes is the time to the first occurrence of all-cause death, liver-related death, liver decompensation, liver transplantation, or hepatocellular carcinoma. All first occurrences were to be included, regardless of whether it occurred while the participant was still taking study drug or had previously discontinued study drug. If the participant did not experience any of these events, their data was to be censored at the date of their last available assessment of clinical outcomes. For participants with no post-baseline assessment, the participant's data was to be censored on the first day of study drug dosing. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. Pre-specified analysis included pooled data from this study and from TOPAZ-I; NCT02219490.
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 11.4 [5.2 to 24.2] | 0.5 [0.3 to 0.9]
  Kaplan-Meier estimate at PT Week 104 | 11.4 [5.2 to 24.2] | 1.2 [0.8 to 1.8]
  Kaplan-Meier estimate at PT Week 156 | 11.4 [5.2 to 24.2] | 1.9 [1.4 to 2.6]
  Kaplan-Meier estimate at PT Week 208 | 11.4 [5.2 to 24.2] | 2.3 [1.7 to 3.1]
  Kaplan-Meier estimate at PT Week 260 | 11.4 [5.2 to 24.2] | 3.2 [2.5 to 4.1]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cox proportional hazards model; Cox Proportional Hazard Ratio = 0.133, 95% CI 2-sided [0.057 to 0.313] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ) 12 weeks after the last actual dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: ITT-II population: all participants enrolled in this study (M14-222; TOPAZ-II) who received at least one dose of study drug. Flanking imputation, where applicable, was used to impute missing data. After applying flanking imputation, if there was no value in the window but there was an HCV RNA value from a local laboratory present, then it was to be imputed into the SVR window. Otherwise, participants with missing data were counted as failures.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV)
Number analyzed (Participants) | 615
percentage of participants | 95.3 [93.3 to 96.7]

8. Secondary Outcome: Mean Change From Baseline in Short Form 36 Version 2.0 (SF-36 V2) Physical Component Summary (PCS) Score at Post-Treatment Week 12 and Post-Treatment Week 24
Description: The SF-36v2 is a non-disease specific Health Related Quality of Life (HRQoL) instrument with extensive use in multiple disease states. The SF-36v2 instrument comprises 36 total items (questions) targeting a subject's functional health and well-being in 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health) with a recall period of 4 weeks. Domain scores are aggregated into a Physical Component Summary (PCS) score and a Mental Component Summary (MCS) score. SF-36v2 scores for each domain and PCS/MCS range from 0-100: higher scores indicate a better state of health. Positive numbers indicate improvement from baseline.
Time Frame: From Baseline to Post-Treatment Week 12 and Post-Treatment Week 24
Population: ITT-II population: all participants enrolled in this study (M14-222; TOPAZ-II) who received at least one dose of study drug and had both baseline and post-treatment data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Fibrosis Stage F0-F1: Participants in study M14-222 with a baseline fibrosis stage of F0 or F1
- Baseline Fibrosis Stage F2: Participants in study M14-222 with a baseline fibrosis stage of F2
- Baseline Fibrosis Stage F3: Participants in study M14-222 with a baseline fibrosis stage of F3
- Baseline Fibrosis Stage F4: Participants in study M14-222 with a baseline fibrosis stage of F4
Arm/Group | Baseline Fibrosis Stage F0-F1 | Baseline Fibrosis Stage F2 | Baseline Fibrosis Stage F3 | Baseline Fibrosis Stage F4
Number analyzed (Participants) | 291 | 85 | 104 | 106
units on a scale
  At Post-treatment Week 12 | 1.2 (6.33) | 0.0 (6.32) | 1.8 (7.80) | 1.4 (7.54)
  At Post-treatment Week 24: number analyzed (Participants) | 288 | 82 | 103 | 103
  At Post-treatment Week 24 | 1.1 (6.86) | 0.5 (7.47) | 2.3 (8.11) | 1.8 (7.77)
Statistical Analysis 1: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F2; F0-F1 vs F2 at Post-treatment Week 12 The difference between baseline fibrosis stage groups in mean change from baseline was analyzed using ANCOVA with baseline fibrosis stage (F0-F1, F2, F3 and F4) as a factor and baseline patient reported outcomes(PRO) score and SVR12 status as covariates; Test type: Superiority; p = 0.026, ANCOVA; LS Mean Difference = -1.75, 95% CI 2-sided [-3.30 to -0.21], Standard Error of Mean 0.79 — F2 - F0-F1
Statistical Analysis 2: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F3; F0-F1 vs F3 at Post-treatment Week 12 The difference between baseline fibrosis stage groups in mean change from baseline was analyzed using ANCOVA with baseline fibrosis stage (F0-F1, F2, F3 and F4) as a factor and baseline patient reported outcomes(PRO) score and SVR12 status as covariates; Test type: Superiority; p = 0.472, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-1.97 to 0.91], Standard Error of Mean 0.74 — F3 - F0-F1
Statistical Analysis 3: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F4; F0-F1 vs F4 at Post-treatment Week 12 The difference between baseline fibrosis stage groups in mean change from baseline was analyzed using ANCOVA with baseline fibrosis stage (F0-F1, F2, F3 and F4) as a factor and baseline patient reported outcomes(PRO) score and SVR12 status as covariates; Test type: Superiority; p = 0.159, ANCOVA; LS Mean Difference = -1.03, 95% CI 2-sided [-2.47 to 0.40], Standard Error of Mean 0.73 — F4 - F0-F1
Statistical Analysis 4: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F2; F0-F1 vs F2 at Post-treatment Week 24 The difference between baseline fibrosis stage groups in mean change from baseline was analyzed using ANCOVA with baseline fibrosis stage (F0-F1, F2, F3 and F4) as a factor and baseline patient reported outcomes(PRO) score and SVR12 status as covariates; Test type: Superiority; p = 0.125, ANCOVA; LS Mean Difference = -1.30, 95% CI 2-sided [-2.95 to 0.36], Standard Error of Mean 0.84 — F2 - F0-F1
Statistical Analysis 5: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F3; F0-F1 vs F3 at Post-treatment Week 24 The difference between baseline fibrosis stage groups in mean change from baseline was analyzed using ANCOVA with baseline fibrosis stage (F0-F1, F2, F3 and F4) as a factor and baseline patient reported outcomes(PRO) score and SVR12 status as covariates; Test type: Superiority; p = 0.756, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-1.78 to 1.29], Standard Error of Mean 0.78 — F3 - F0-F1
Statistical Analysis 6: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F4; F0-F1 vs F4 at Post-treatment Week 24 The difference between baseline fibrosis stage groups in mean change from baseline was analyzed using ANCOVA with baseline fibrosis stage (F0-F1, F2, F3 and F4) as a factor and baseline patient reported outcomes(PRO) score and SVR12 status as covariates; Test type: Superiority; p = 0.315, ANCOVA; LS Mean Difference = -0.79, 95% CI 2-sided [-2.32 to 0.75], Standard Error of Mean 0.78 — F4 - F0-F1

9. Secondary Outcome: Mean Change From Baseline in Short Form 36 Version 2.0 (SF-36 V2) Mental Component Summary (MCS) Score at Post-Treatment Week 12 and Post-Treatment Week 24
Description: as for outcome 8
Time Frame: From Baseline to Post-Treatment Week 12 and Post-Treatment Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline Fibrosis Stage F0-F1 | Baseline Fibrosis Stage F2 | Baseline Fibrosis Stage F3 | Baseline Fibrosis Stage F4
Number analyzed (Participants) | 291 | 85 | 104 | 106
units on a scale
  At Post-treatment Week 12 | 2.7 (9.77) | 1.0 (9.05) | 0.9 (9.64) | 0.3 (10.62)
  At Post-treatment Week 24: number analyzed (Participants) | 288 | 82 | 103 | 103
  At Post-treatment Week 24 | 3.2 (9.85) | 1.9 (7.28) | 1.5 (10.73) | 0.4 (10.20)
Statistical Analysis 1: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F2; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.216, ANCOVA; LS Mean Difference = -1.28, 95% CI 2-sided [-3.30 to 0.75], Standard Error of Mean 1.03 — F2 - F0-F1
Statistical Analysis 2: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F3; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = 0.074, ANCOVA; LS Mean Difference = -1.70, 95% CI 2-sided [-3.58 to 0.17], Standard Error of Mean 0.95 — F3 - F0-F1
Statistical Analysis 3: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F4; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.056, ANCOVA; LS Mean Difference = -1.81, 95% CI 2-sided [-3.67 to 0.05], Standard Error of Mean 0.95 — F4 - F0-F1
Statistical Analysis 4: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F2; [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p = 0.411, ANCOVA; LS Mean Difference = -0.84, 95% CI 2-sided [-2.84 to 1.16], Standard Error of Mean 1.02 — F2 - F0-F1
Statistical Analysis 5: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F3; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.065, ANCOVA; LS Mean Difference = -1.72, 95% CI 2-sided [-3.55 to 0.11], Standard Error of Mean 0.93 — F3 - F0-F1
Statistical Analysis 6: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F4; F0-F1 vs F4 at Post-treatment Week 24; Test type: Superiority; p = 0.026, ANCOVA; LS Mean Difference = -2.08, 95% CI 2-sided [-3.91 to -0.25], Standard Error of Mean 0.93 — F4 - F0-F1

10. Secondary Outcome: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Total Score at Post-Treatment Week 12 and Post-Treatment Week 24
Description: The FACIT-F is a symptom specific instrument with a focus on measuring fatigue in a variety of chronic diseases or health conditions. It was originally developed from interviews with oncology patients and clinical experts to assess anemia-associated fatigue. Its 13-item-version assesses peripheral, central, or mixed fatigue with a recall period of 7 days and yields a summed total score ranging between 0 and 52. Higher FACIT-F scores indicate a lesser degree of fatigue. Positive numbers indicate improvement from baseline.
Time Frame: From Baseline to Post-Treatment Week 12 and Post-Treatment Week 24
Population: ITT-II population: all participants enrolled in this study (M14-222; TOPAZ-II) who received at least one dose of study drug who had both baseline and post-treatment data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline Fibrosis Stage F0-F1 | Baseline Fibrosis Stage F2 | Baseline Fibrosis Stage F3 | Baseline Fibrosis Stage F4
Number analyzed (Participants) | 292 | 86 | 103 | 105
units on a scale
  At Post-treatment Week 12 | 3.9 (9.66) | 2.0 (9.12) | 2.0 (8.63) | 3.0 (9.57)
  At Post-treatment Week 24: number analyzed (Participants) | 289 | 82 | 103 | 103
  At Post-treatment Week 24 | 3.9 (10.46) | 3.1 (6.85) | 2.3 (9.27) | 2.6 (10.88)
Statistical Analysis 1: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F2; F0-F1 vs F2 at Post-treatment Week 12 The difference between baseline fibrosis stage groups in mean change from baseline was analyzed using ANCOVA with baseline fibrosis stage (F0-F1, F2, F3 and F4) as a factor and baseline patient reported outcomes (PRO) score and SVR12 status as covariates; Test type: Superiority; p = 0.035, ANCOVA; LS Mean Difference = -2.00, 95% CI 2-sided [-3.86 to -0.14], Standard Error of Mean 0.95 — F2 - F0-F1
Statistical Analysis 2: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F3; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = 0.015, ANCOVA; LS Mean Difference = -2.15, 95% CI 2-sided [-3.88 to -0.42], Standard Error of Mean 0.88 — F3 - F0-F1
Statistical Analysis 3: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F4; F0-F1 vs F4 at Post-treatment Week 12; Test type: Superiority; p = 0.048, ANCOVA; LS Mean Difference = -1.74, 95% CI 2-sided [-3.46 to -0.01], Standard Error of Mean 0.88 — F4 - F0-F1
Statistical Analysis 4: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F2; [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p = 0.466, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-2.67 to 1.22], Standard Error of Mean 0.99 — F2 - F0-F1
Statistical Analysis 5: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F3; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.035, ANCOVA; LS Mean Difference = -1.91, 95% CI 2-sided [-3.70 to -0.13], Standard Error of Mean 0.91 — F3 - F0-F1
Statistical Analysis 6: Comparison: Baseline Fibrosis Stage F0-F1 vs Baseline Fibrosis Stage F4; [analysis description as in outcome 8, analysis 6]; Test type: Superiority; p = 0.015, ANCOVA; LS Mean Difference = -2.22, 95% CI 2-sided [-4.01 to -0.43], Standard Error of Mean 0.91 — F4 - F0-F1

11. Secondary Outcome: Treatment Compliance: Percentage of Tablets Taken Relative to the Total Tablets
Description: Treatment compliance was calculated as the percentage of tablets taken (presumed as [tablets dispensed-tablets returned]) relative to the total tablets, respectively, expected to be taken. Study drug interruptions due to an adverse event or other planned interruptions recorded on the electronic case report form (eCRF) were to be subtracted from the duration. For compliance to ribavirin (RBV), RBV dose modifications due to adverse events, toxicity management, or weight changes as recorded on the RBV Dose Modifications eCRF were to be used to modify the total number of tablets that should have been taken. A participant is considered to be compliant if the percentage is between 80% and 120%.
Time Frame: Up to Treatment Week 24
Population: Safety population: all participants enrolled in this study (M14-222; TOPAZ-II) who received at least one dose of study drug with available data
Measure: Mean (Standard Deviation); unit: percentage of tablets taken
Groups:
- ABT-450/r/ABT-267 Plus ABT-333: Participants with HCV GT1b without cirrhosis received the 3-DAA (ABT-450/ritonavir/ABT-267 and ABT-333) regimen: two 75 mg ABT-450/50 mg ritonavir/12.5 mg ABT-267 tablets taken orally every morning (QD) and one ABT-333 250 mg tablet taken orally twice a day (BID) for 12 weeks. Participants with HCV GT1a without cirrhosis and those with HCV GT1b with cirrhosis received the 3-DAA regimen for 12 weeks. Participants with HCV GT1a with cirrhosis received the 3-DAA regimen for 24 weeks.
- Weight-based Ribavirin (RBV): Participants with HCV GT1a without cirrhosis and those with HCV GT1b with cirrhosis received weight-based ribavirin (RBV; 1000 to 1200 mg divided twice daily per local label) for 12 weeks. Participants with HCV GT1a with cirrhosis received weight-based RBV per local label for 24 weeks. Ribavirin was provided as 200 mg tablets, and dosed based on weight, 1000 to 1200 mg divided twice daily per local label. For example, for participants weighing < 75 kg, RBV may have been taken orally as 2 tablets in the morning and 3 tablets in the evening which corresponds to a 1000 mg total daily dose. For participants weighing ≥ 75 kg, RBV may have been taken orally as 3 tablets in the morning and 3 tablets in the evening which corresponds to a 1200 mg total daily dose.
Arm/Group | ABT-450/r/ABT-267 Plus ABT-333 | Weight-based Ribavirin (RBV)
Number analyzed (Participants) | 567 | 408
percentage of tablets taken | 100.22 (22.88) | 99.86 (12.40)

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to the end of study, up to five years of follow-up. Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 30 days after the last study drug administration, up to 213 days. After Post-Treatment Week 4 until the end of the study, only SAE of death was to be collected.
Description: All-cause mortality and adverse events: all participants in this study (M14-222; TOPAZ-II) who received at least one dose of study drug
Arm/Group | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV)
All-Cause Mortality (participants affected / at risk) | 19/615
Serious Adverse Events (participants affected / at risk) | 25/615
Other Adverse Events (participants affected / at risk) | 381/615
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV) (N=615)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1)
PERICARDITIS (Cardiac disorders) | 1 (1)
HYPERADRENOCORTICISM (Endocrine disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
CHEST PAIN (General disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
ALLERGIC OEDEMA (Immune system disorders) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
PERITONITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 2 (2)
SCHIZOAFFECTIVE DISORDER (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV) (N=615)
ANAEMIA (Blood and lymphatic system disorders) | 32 (32)
DIARRHOEA (Gastrointestinal disorders) | 54 (59)
NAUSEA (Gastrointestinal disorders) | 99 (104)
VOMITING (Gastrointestinal disorders) | 31 (32)
FATIGUE (General disorders) | 198 (209)
DIZZINESS (Nervous system disorders) | 37 (38)
HEADACHE (Nervous system disorders) | 98 (101)
INSOMNIA (Psychiatric disorders) | 78 (80)
COUGH (Respiratory, thoracic and mediastinal disorders) | 35 (35)
PRURITUS (Skin and subcutaneous tissue disorders) | 87 (89)
RASH (Skin and subcutaneous tissue disorders) | 49 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2014-12-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT02167945/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT02167945/SAP_001.pdf